CLINICAL TRIAL: NCT06077266
Title: Factors Associated With Changes in Weight-status in Danish School Children: From Obesity to Overweight or Normal Weight
Brief Title: Factors Associated With Changes in Weight-status in Danish School Children With Obesity
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Municipality, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: Journal no.: 2022-0367531
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Obesity
Keywords: Weight Loss; Body-Weight Trajectory
MeSH Terms: conditions — Pediatric Obesity; Weight Loss; Body-Weight Trajectory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normalizing weight: Children classified as having normalized weight (iso-BMI 18.5-25 for age and sex) at the last observation defined by IOTF.
  Interventions: Other: Change of weight class to normal weight
- Overweight or obesity: Children classified as having overweight or obesity (iso-BMI 25 ≤ for age and sex) at the last observation defined by IOTF.

INTERVENTIONS:
Other: Change of weight class to normal weight — The exposure is the change of weight class from obesity to normal weight during a follow-up period without known intervention.
  Groups: Normalizing weight

SUMMARY:
Childhood obesity is increasing worldwide and causes a major health concern. Only limited insight exists into the natural history of childhood obesity at children already classified as obese. It is necessary to identify possible windows of opportunities to initiate treatment and to prevent further weight gain later in life.

This observational study follows the natural weight change in younger children with obesity without known intervention. The objective is to identify factors associated with achieving normal weight, having persistent obesity, or reaching higher levels of obesity, when following children age 5-10 years with obesity through childhood and puberty.

Data from health check-ups at school and Danish registries will be used to answer the research question.

DETAILED DESCRIPTION:
Only limited insight exists into the natural history of childhood obesity at children already classified as obese. It is necessary to identify possible windows of opportunities to initiate treatment and to prevent further weight gain later in life.

High Body Mass Index (BMI) or weight status early in life seems to predict the risk of persisting obesity and indicating BMI as an important predictor for the chance of remission. High birthweight has also been associated with poor chance of normalizing weight, when following children with obesity from kindergarten to the 8th grade, indicating that severe obesity can be detectable from early childhood.

Children with severe obesity (iso-BMI ≥ 35) have been observed to gain weight with a faster rate and with a critical period between 12 to 14 years of age, compared to children with less-severe obesity (iso-BMI < 35). Another report observes, that having obesity at the age of six was associated with obesity after puberty, while no such association was observed for younger children (six years). Hereby suggesting that children at a younger age have chance of achieving remission of obesity, than children classified as having obesity later in life.

Other factors such as sex, ethnicity and interpersonal skills have also been observed to influence the chance of normalizing weight, when following children with obesity from 5th to 8th grade.

This study aims to identify factors associated with achieving normal weight, when following children age 5-10 yrs. with obesity through childhood and puberty.

In addition, to identify factors associated with having persisting obesity, or reaching a higher level of obesity (highest 20% increase in BMI z-score from baseline)

The participants:

This study includes Danish children 5 to 10 years of age with obesity with minimum three years of follow-up during. Children invited into the local community-based lifestyle intervention will be excluded. The IOTF cut-offs for weight status at the last obtained observation will be used to define the groups.

Data sources:

1. Observations containing anthropometrics have been extracted from TM-Sund for each child. TM-Sund is a database used in Aarhus municipality to store data on anthropomet-rics obtained at health checks at the school (read more on https://www.solteq.com/da).
2. Data on family structure, socioeconomic status (SES), immigration status and psychiatric diagnoses (child and parents) will be obtained from Danish registries at Statistics Den-mark.
3. The local registry at Aarhus Municipality will be used to identify and exclude children 1) treated in or 2) declined participation in a lifestyle intervention.

Statistics:

A logistic regression analysis will be used to identify baseline factors associated with the group of children normalizing weight, persistent obesity and highest increase of BMI z-score (above the 20th centile) at the last observation, respectively. Observations will be weighted by the possible follow-up.

Ethics & permissions:

The Danish Data Protection Agency and the local committee on health ethics have approved the overall project and data transfer (rec.no 1-45-70-27-2).

ELIGIBILITY:
Inclusion Criteria:

1. Baseline visit between January 1st. 2010 and March 17th 2018.
2. Minimum one observation with obesity
3. Minimum three years of follow-up from baseline
4. Children age 5-10 years

Exclusion Criteria:

1. Children registered in a community-based lifestyle intervention.
2. Children registered as having declined participation in a community-based lifestyle intervention.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population consist of children with obesity from the city of Aarhus, Denmark between January 1st 2010 and March 18nd 2018, but followed until March 18nd 2021.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Factors associated with changes in weight-status in Danish school children: from obesity to normal weight. | Children with a baseline visit between January the 1st 2010 and March the 18nd 2018 will be included. The children will be followed until March the 18nd 2021.
  Factors associated with changes in weight-status in Danish school children (age 5-10 years) from obesity or normal weight. Only children with minimum 3 years of follow-up will be included.
  Children treated in or declining treatment in a lifestyle intervention for obesity will be excluded.

SECONDARY OUTCOMES:
Factors associated with persisting obesity in Danish school children with obese. | Children with a baseline visit between January the 1st 2010 and March the 18nd 2018 will be included. The children will be followed until March the 18nd 2021.
  Factors associated persisting obesity in Danish school children (age 5-10 years) compared to children obtaining remission of obesity. Only children with obesity at baseline and minimum 3 years of follow-up will be included. Children treated in or declining treatment in a lifestyle intervention for obesity will be excluded.
Factors associated with the highest increase in BMI z-score (above the 20th percentile) in Danish school children with obese. | Children with a baseline visit between January the 1st 2010 and March the 18nd 2018 will be included. The children will be followed until March the 18nd 2021.
  Factors associated the highest increase in BMI z-score (above the 20th percentile in changes from baseline) in Danish school children (age 5-10 years) compared to children with lower increase or decrease in BMI z-score (below the 20th percentile within the cohort). Only children with minimum 3 years of follow-up will be included. Children treated in or declining treatment in a lifestyle intervention for obesity will be excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data can be shared upon publication on a reasonable request. However, data from the National registries cannot be shared due to Danish General Data Protection Regulation and legislation.